CLINICAL TRIAL: NCT04083495
Title: Phase II Study of the Administration of T Lymphocytes Expressing the CD30 Chimeric Antigen Receptor (CAR) for Relapsed/Refractory CD30+ Peripheral T Cell Lymphoma
Brief Title: CD30 CAR for Relapsed/Refractory CD30+ T Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1904-ATL
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: lymphoma; CD30; peripheral T cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma | interventions — Bendamustine Hydrochloride; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATLCAR.CD30 cells (Experimental): The cellular product consisting of ATLCAR.CD30 cells will be administered via intravenous injection over 5 - 10 minutes through either a peripheral or a central line. The volume of infusion will depend upon the concentration of the cells when frozen and the size of the subject. Administration to eligible subjects will occur within 2 - 14 days after completing the lymphodepleting chemotherapy regimen
  Interventions: Biological: ATLCAR.CD30 T cells; Drug: Bendamustine; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: ATLCAR.CD30 T cells — Autologous T Lymphocyte Chimeric Antigen Receptor cells targeted against the CD30 antigen at dose of 2 × 10^8 CAR-T/m^2 with a maximum dose of 5 × 10^8 CAR-T cells
Drug: Bendamustine — 70 mg/m^2 administered IV for 3 days for lymphodepletion 2-14 days prior to first cell infusion
  Other Names: Bendeka
Drug: Fludarabine — 30 mg/m^2 administered IV for 3 days for lymphodepletion 2-14 days prior to first and second cell infusion
Drug: Cyclophosphamide — 300 mg/m^2 administered IV for 3 days for lymphodepletion 2-14 days prior to second cell infusion and 2-14 days prior to the first cell infusion for subjects who have previously had hypersensitivity to bendamustine

SUMMARY:
This is a research study to determine the safety and tolerability of ATLCAR.CD30 for treating relapsed/refractory Peripheral T Cell Lymphoma. Blood samples will be collected from study participants and the immune T cells will be separated. T cells will be genetically modified in a laboratory at UNC-Chapel Hill to enable them to produce CD30 antibody. The modified T cells, called ATLCAR.CD30, will be able to target and attach to lymphoma cancer cells that carry the CD30 antigen. Once they are attached, the hope is that the T cells will attack and destroy the lymphoma cancer cells. To prepare the body for the ATLCAR.CD30 cells, participants will complete lymphodepletion with two chemotherapy agents. Lymphodepletion will happen over three days prior to ATLCAR.CD30 infusion. If participants respond to this treatment, and there are sufficient unused ATLCAR.CD 30 cells, they may be eligible to receive a second infusion. The second infusion will be given after a second lymphodepletion chemotherapy. Most of the clinic visits in this research will last between 1-8 hours.

There are risks associated in participating in this research study. Risks of treatment include infection, fever, nausea, vomiting, neurotoxicity, and cytokine release syndrome which can include low blood pressure or difficulty breathing. Other risks are associated with study procedures, such as biopsies, imaging, infusion, and breach of confidentiality.

DETAILED DESCRIPTION:
This multicenter, open-label phase II study will determine the efficacy and safety of autologous activated T lymphocytes (ATLs) expressing the chimeric antigen receptor specific for CD30 (ATLCAR.CD30) administered in two sequential infusions in subjects with relapsed/refractory CD30+ PTCL. Up to 20 subjects will receive 2 infusions of 2 × 108 cells/m2 of ATL product expressing the CAR.CD30. It can take time to procure the subjects cells and manufacture the ATLCAR.CD30 cells. During the time period required to manufacture the product the subjects will be able to receive standard of care bridging therapy to be determined by their primary local oncologist. Prior to receiving the first cell infusion, subjects will undergo lymphodepletion with fludarabine and bendamustine. Any subject with prior hypersensitivity reaction to bendamustine will be considered for an alternative lymphodepletion regimen. Subjects will have their disease assessed at week 8 by either CT chest, abdomen and pelvis or PET/CT. Subjects who have stable disease (SD), partial response (PR) or complete response (CR) without subsequent progressive disease and meet the eligibility criteria for a second infusion, will receive lymphodepletion followed by a second infusion. The lymphodepletion for the second infusion will consist of cyclophosphamide and fludarabine.

OUTLINE

Cell Procurement Up to 300 mL of peripheral blood (in up to 3 collections) will be obtained from subjects for cell procurement. Additionally, leukapheresis may be performed to isolate sufficient cells in subjects with a low absolute lymphocyte count or who had inadequate peripheral blood collection. The parameters for apheresis will be up to 2 blood volumes.

Bridging Chemotherapy while waiting for CAR_T cells to be prepared Subjects will be allowed to receive additional standard of care therapy (e.g., chemotherapy or radiation therapy) to stabilize their disease if the treating physician feels it is in the subject's best interests.

Lymphodepleting Chemotherapy Prior to the initial cellular product administration subjects will receive a lymphodepleting regimen of bendamustine 70 mg/m^2/day administered IV over 1 hour followed by an IV dose over 30 minutes of fludarabine 30 mg/m^2/day administered over 3 consecutive days. These agents will be administered per institutional guidelines. Prophylaxis (e.g., hydration, antiemetics, etc.) needed prior to fludarabine and bendamustine chemotherapy will be provided per institutional guidelines. Lymphodepletion will be given 2-14 days prior to the initial cell product administration. Subjects who have previously had hypersensitivity to bendamustine may receive a lymphodepletion regimen of cyclophosphamide 300 mg/m^2 IV and fludarabine 30 mg/m^2 each as a daily infusion for 3 days 2-14 days prior to the initial cell product administration.

Two to 14 days prior to the second infusion, subjects will receive a lymphodepletion regimen of cyclophosphamide 300 mg/m^2 IV and fludarabine 30 mg/m^2 each as a daily infusion for 3 days per institutional guidelines. Subjects whose absolute neutrophil count and/or platelet count takes >/= 3 months (from the first day of lymphodepletion prior to the initial cellular product administration) to recover to levels required to meet eligibility for lymphodepletion (ANC >/= 1.0 x 10^9/L and platelet count >/= 50 x 10^9/L) prior to the second infusion will receive a 25% dose reduction in cyclophosphamide and fludarabine lymphodepletion for the second round of lymphodepletion.

ATLCAR.CD30 Cell Administration The cellular product consisting of ATLCAR.CD30 cells will be administered by a licensed healthcare provider (oncology nurse or physician) via intravenous injection over 5 - 10 minutes through either a peripheral or a central line. The volume of infusion will depend upon the concentration of the cells when frozen and the size of the subject. The expected volume will be 1 - 50 mL. Post lymphodepletion, subjects who meet eligibility criteria for cellular therapy will receive ATLCAR.CD30 cells within 2 - 14 days after completing the lymphodepleting chemotherapy regimen. The recommended phase 2 dose (RP2D) determined in the phase 1 study of ATLCAR.CD30 will be administered to subjects (2 × 108 CAR-T/m2).

If a subject only has enough ATLCAR.CD30 cells product for one infusion, they will still be able to receive one infusion of cells and will not have a 2nd lymphodepletion or infusion of cells. These subjects will be replaced for the purposes of efficacy determination.

Duration of Therapy

Therapy in the study involves 2 infusions of ATLCAR.CD30 cells. Treatment with at least one infusion will be administered unless:

* Subject decides to withdraw from study treatment, or
* General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator.

Duration of Follow-Up

* Subjects will be followed for up to 15 years from final cell product administration or until death, whichever occurs first.
* Subjects removed from study treatment for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.
* Subjects who experience unequivocal disease progression and start alternate therapy after receiving a cell infusion will still be required to complete abbreviated follow up procedures outlined in the protocol.

ELIGIBILITY:
Inclusion Criteria for the Study

1. Written informed consent and HIPAA authorization for release of personal health information explained to, understood by and signed by the subject or legally authorized representative.
2. Age ≥ 18 years at the time of consent.
3. Karnofsky score of >60%
4. Histological or cytological evidence/confirmation of CD30+ peripheral T-cell lymphoma per the 2017 World Health Organization Classification of Haematopoietic and Lymphoid Tissues.
5. CD30+ disease determined via archival tissue after the subject's most recent anti-CD30 therapy prior to ATLCAR.CD30 (result can be pending at the time of cell procurement but must be confirmed prior to treatment with the first infusion of ATLCAR.CD30 cells). NOTE: CD30+ disease requires documented CD30 expression by immunohistochemistry based on the institutional hematopathology standard.
6. Any subjects who has received at least two prior lines of therapy for their lymphoma. If transplant is given as a preplanned consolidation in first remission, it will not be counted as a second line of therapy.
7. Any subject who has received one line of therapy who has primary refractory lymphoma or lymphoma that relapsed within 12 months of completing chemotherapy or receiving transplant as long as prior therapy included brentuximab vedotin unless they were not candidates for brentuximab vedotin.
8. Subjects relapsed after autologous stem cell transplant are eligible for this study.
9. Subjects relapsed after allogeneic stem cell transplantation are eligible provided the patient is ≥180 days from transplant, not on immunosuppresive therapy to treat/prevent graft-versus-host disease and has no evidence of active graft-versus-host disease.
10. Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
11. Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to cell procurement. Note: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided.
12. Female subjects of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 6 months after study treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets <1% failure rate for protection from pregnancy in the product label. Women of childbearing potential will also be instructed to tell their male partners to use a condom.
13. Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.

Exclusion Criteria for the Study

1. Subject is pregnant or lactating (Note: Breast milk cannot be stored for future use while the mother is being treated on study ).
2. Current use of systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent; those receiving <10 mg daily may be enrolled at discretion of investigator. Inhaled steroids are allowed.
3. Active infection with HIV, HTLV, HCV (tests can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells). Note: To meet eligibility subjects are required to be negative for HIV antibody, negative for HTLV1 and 2 antibody or PCR negative for HTLV1 and 2, negative for HCV antibody or HCV viral load.
4. Subjects who are positive for hepatitis B surface antigen (can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells) are excluded. Subjects who are hepatitis B surface antigen negative but hepatitis B core antibody positive must have their hepatitis B viral load checked. These subjects will be excluded if their viral load is positive at baseline. Subjects who are core antibody positive and viral load negative at baseline will be considered eligible.

Eligibility Criteria Prior to Cell Procurement

1. Informed consent to undergo cell procurement understood by and signed by the subject or legally authorized representative; subject and/or legally authorized representative given a copy of informed consent form for cell procurement.
2. Subject has life expectancy ≥ 6 weeks.
3. Subject has evidence of adequate organ function within 7 days of procurement as defined by:

   * Hemoglobin ≥8.0 g/dL (transfusion is allowed prior to procurement)
   * Total bilirubin ≤ 2 × ULN, unless attributed to Gilbert's Syndrome
   * AST ≤ 3 × ULN
   * ALT < 3 x ULN
   * Creatinine ≤ 2 × ULN
   * Pulse oximetry of >90% on room air
4. Imaging results from within 90 days prior to procurement to assess presence of active disease.
5. Negative serum pregnancy test within 72 hours prior to procurement or documentation that the subject is post-menopausal. Post-menopausal status must be confirmed with documentation of absence of menses for >1 year, or documentation of surgical menopause (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.

Eligibility Criteria Prior to Lymphodepletion #1

1. Written informed consent explained to, understood by and signed by the subject or legally authorized representative; subject and/or legally authorized representative given a copy of informed consent form.
2. Imaging results from within 10 days prior to lymphodepletion. Imaging must occur at least 3 weeks after most recent therapy (used as baseline measure for documentation of progression before the lymphodepletion) to document measurable or assessable disease.
3. Subject must demonstrate adequate organ function prior to lymphodepletion as defined below. All tests must be obtained within 72 hours prior to lymphodepletion:

   * Absolute neutrophil count ≥ 1.0 × 10^9/L
   * Platelet count ≥ 50 × 10^9/L
   * Total bilirubin < 2 x ULN unless attributed to Gilbert's syndrome
   * AST ≤ 5 x ULN
   * ALT ≤ 5 x ULN
   * Creatinine ≤ 3 x ULN
   * Pulse Oximetry of >90% on room air
4. Subject must have available autologous transduced activated T cells product at a dose of 2x10^8 cells/m^2 and meets the Certificate of Analysis acceptance criteria.
5. No major surgery within 28 days prior to lymphodepletion.
6. Negative serum pregnancy test within 72 hours prior to lymphodepleting therapy for female participants of childbearing potential. Note: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
7. Subject has not received any investigational agents or any tumor vaccines within the previous six weeks prior to lymphodepletion.
8. Subject has not received anti-CD30 antibody-based therapy within the previous 4 weeks prior to lymphodepletion.
9. Subject has not received chemotherapy within the previous 3 weeks prior to lymphodepletion.
10. Subject does not have rapidly progressive disease, per treating oncologist's discretion.
11. Subject is a good candidate for CAR T cell therapy, per treating oncologist's discretion.
12. Subjects on strong inhibitors of CYP1A2 (e.g., fluvoxamine, ciprofloxacin) as these may increase plasma concentrations of bendamustine, and decrease plasma concentrations of its metabolites. See http://medicine.iupui.edu/clinpharm/ddis/ for an updated list of strong inhibitors of CYP1A2. (This applies to subjects who receive bendamustine for lymphodepletion (required) up through 72 hours after the last dose of bendamustine.)
13. Subject is not taking a prohibited or contraindicated medication prior to lymphodepletion.
14. Current use of systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent; those receiving <10 mg daily may be enrolled at discretion of investigator. Inhaled steroids are allowed.

Eligibility Criteria Prior to Cell Product Administration #1

1. Subject has no evidence of uncontrolled infection or sepsis.
2. Negative serum pregnancy within 7 days of cell product administration for females of childbearing potential (does not need to be repeated if pre-lymphodepletion pregnancy test is within window). Note: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oopherectomy) or they are naturally postmenopausal for at least 12 consecutive months.
3. Evidence of adequate organ function as defined by:

   * Total bilirubin ≤ 2 × ULN, unless attributed to Gilbert's syndrome
   * AST ≤ 5 × ULN
   * ALT ≤ 5 × ULN
   * Creatinine ≤ 3 × ULN
   * Pulse Oximetry of >90% on room air
4. Subject has no clinical indication of rapidly progressing disease in the opinion of the clinical investigator.
5. Subject is a good candidate for treatment with ATLCAR.CD30 cell product per the clinical investigator's discretion.

Eligibility Criteria Prior to Lymphodepletion #2

1. Imaging results from within 21 days prior to lymphodepletion to confirm that the subject has derived clinical benefit from the initial infusion as assessed by the investigator. Clinical benefit will be defined as:

   1. Subject with stable disease or better after the first ATLCAR.CD30 infusion without subsequent progressive disease.
   2. Subjects that had a PR or CR and progressed after the first ATLCAR 30 infusion and prior to second lymphodepletion. A second infusion will be made available to the subject, if the subject chooses, if the treating investigator suspects the subject would obtain clinical benefit from a second infusion and all other eligibility criteria are met.
2. Subjects who experienced Grade 4 CRS or Grade 4 ICANS as a result of the initial ATLCAR.CD30 infusion are only eligible for a second round of lymphodepletion and infusion if they have partial response or better to the initial ATLCAR.CD30 infusion.
3. Subject must demonstrate adequate organ function prior to lymphodepletion as defined below. All tests must be obtained within 24 hours prior to lymphodepletion:

   * Absolute neutrophil count ≥ 1.0 × 10^9/L
   * Platelet count ≥ 50 × 10^9/L
   * Total bilirubin ≤ 2 × ULN, unless attributed to Gilbert's syndrome
   * AST ≤ 5 × ULN
   * ALT ≤ 5 × ULN
   * Creatinine ≤ 3 × ULN
   * Pulse Oximetry of >90% on room air
4. Subject must have available autologous transduced activated T cells product at a dose of 2x10^8 cells/m^2 and meets the Certificate of Analysis acceptance criteria.
5. Negative serum pregnancy test within 72 hours prior to lymphodepleting therapy for female participants of childbearing potential. Note: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
6. Subject does not have evidence of uncontrolled infection or sepsis.
7. Subject is not receiving a prohibited medication at time of starting lymphodepletion up through 72 hours after the last dose of cyclophosphamide.
8. Subject is a good candidate for CAR T cell therapy, per treating oncologist's discretion.
9. Current use of systemic corticosteroids at doses ≥10 mg prednisone daily or its equivalent; those receiving <10 mg daily may be enrolled at discretion of investigator. Inhaled steroids are allowed.

Eligibility Criteria Prior to Cell Product Administration #2

1. Subject has no evidence of uncontrolled infection or sepsis.
2. Negative serum pregnancy within 7 days of cell product administration for females of childbearing potential (does not need to be repeated if pre-lymphodepletion pregnancy test is within window). Note: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
3. Evidence of adequate organ function as defined by:

   * Total bilirubin ≤ 2 × ULN, unless attributed to Gilbert's syndrome
   * AST ≤ 5 × ULN
   * ALT ≤ 5 × ULN
   * Creatinine ≤ 3 × ULN
   * Pulse Oximetry of >90% on room air
4. Subject has no clinical indication of rapidly progressing disease in the opinion of the clinical investigator.
5. Subject is a good candidate for treatment with ATLCAR.CD30 cell product per the clinical investigator's discretion.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2028-02-23 (Estimated); Study Completion 2038-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) after administration of the ATLCAR.CD30 in subjects with relapsed/refractory CD30+ peripheral T cell lymphoma | 8 weeks
  PFS is defined from day of initial lymphodepletion administration of the first ATLCAR.CD30 product infusion to the date of disease progression per the Revised Lugano Criteria or death as a result of any cause. Subjects who do not meet criteria for progression by the analysis data cut-off date will be censored at their last evaluable disease assessment date.

SECONDARY OUTCOMES:
Best overall response rate (BOR) mediated by the ATLCAR.CD30 product administered in subjects with relapsed/refractory CD30+ peripheral T cell lymphoma | 2 years
  The best overall response rate (BOR) will be defined as the best response recorded from the first administration of the ATLCAR.CD30 product to the date of disease progression per the Revised Lugano Criteria or death as a result of any cause.
Objective response rate (ORR) mediated by the first infusion of the ATLCAR.CD30 product administered in patients with relapsed/refractory CD30+ peripheral T cell lymphoma. | 8 weeks
  The objective response rate (ORR) will be defined as the rate of complete responses (CR) + partial responses (PR) by 8 weeks from the date of first lymphodepletion prior to the first administration of the ATLCAR.CD30 product per the Revised Lugano Criteria.
Responses improved by the second infusion of the ATLCAR.CD30 product administered in subjects with either partial response or stable disease following the first infusion of ATLCAR.CD30 | 8 weeks
  The percentage of subjects who have an improvement in their response after the second administration of ATLCAR.CD30 product will be defined at 8 weeks after the second administration of the ATLCAR.CD30 product per the Revised Lugano Criteria. Subjects entering the second infusion in a complete response will be reported as continued CR (CCR) but will not be included in percentage of improved responses after the second infusion.
Incidence of Dose Limiting Toxicity (DLT) (safety and tolerability) when administering two sequential infusions of the ATLCAR.CD30 product in subjects with relapsed/refractory CD30+ peripheral T cell lymphoma | 8 weeks
  DLT defined as ≥ Grade 3 cytokine release syndrome (CRS), Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS), or any other ≥ Grade 3 non-hematologic toxicity, including allergic reactions to T cell infusions. Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. CRS toxicity will be graded according to CRS Grading Criteria and Management Guidelines Version 3.0 (March 14, 2019). ICANS toxicity will be graded according to the ICANS Grading Criteria for Management of Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) for CAR T-Cell Therapy.
Overall survival (OS) after administration of the ATLCAR.CD30 administered to subjects with relapsed/refractory CD30+ peripheral T cell lymphoma | 15 years
  Overall survival is defined from day of initial lymphodepletion for the first administration ATLCAR.CD30 product to date of death.
Comparison of the expansion and persistence of ATLCAR.CD30 in peripheral blood when infused after a single infusion of ATLCAR.CD30 cells and after two infusions with ATLCAR.CD30 cells | 1 year
  Persistence and expansion of ATLCAR.CD30 in peripheral blood after a single infusion and after two infusions will be determined by quantitative polymerase chain reaction (PCR) and flow cytometry in sample of peripheral blood. Feasibility is defined as ability of subjects to receive 2 sequential infusions taking into account manufacturing and any other limiting factors to receiving a second infusion of ATLCAR.CD30

CONTACTS AND LOCATIONS:
Overall Officials: Anne Beaven, MD, Principal Investigator — UNC Chapel Hill
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — https://unclineberger.org/